CLINICAL TRIAL: NCT01563796
Title: A Multi-Center Study to Evaluate the Safety and Efficacy of a Urine DEK ELISA in Diagnosis of Subjects With Bladder Cancer
Brief Title: Efficacy Study of a Urine DEK ELISA for Diagnosis of Bladder Cancer
Status: Terminated | Type: Observational
Why Stopped: Business decision made not to pursue malignant disease diagnostic devices
Sponsor: Medical Diagnostic Laboratories, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ONC04
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hematuria; Dysuria; Bladder Cancer
Keywords: bladder cancer; TCC; urine; protein ELISA
MeSH Terms: conditions — Hematuria; Dysuria; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TCC positive: subjects with hematuria, dysuria or other irritative voiding symptoms, without evidence of other causative factors such as infections or stones that are found to have a bladder tumor confirmed by histopathology
- TCC negative: subjects with hematuria, dysuria or other irritative voiding symptoms, without evidence of other causative factors such as infections or stones that are found to NOT have a bladder tumor by histopathology or clinical observation.

SUMMARY:
The objective of this study is to use a DEK ELISA to quantitatively measure DEK protein in the urine of patients suspected of having bladder cancer. The measurement of urine DEK protein, relative to an established cut-off, is correlated with the presence or absence of bladder cancer.

DETAILED DESCRIPTION:
Sample Collection:

Urine samples used in the study will be collected immediately prior to the urological evaluation procedure and stored at -80 oC. Urine samples will be sent to sponsor and remain at -80o C until analysis.

Clinical Data Collection:

All subject and clinical information will be recorded on the form in section 9.3. Enrollment Checklist and Case Report Form (CRF). Information regarding the history of hematuria and urine cytology will be recorded. In addition, non-identifying information including age, sex, race, smoking history, alcohol consumption, occupational exposure to chemicals or dyes, history of urologic disorder or disease, history of irritative voiding symptoms, history of urinary tract infection, history of pelvic irradiation, and analgesic abuse will be recorded. The Investigators will also be asked to provide information from the subjects' medical records for up to one (1) year after their enrollment and sample collection. In particular, diagnosis of TCC, other malignant diseases, or non-malignant urogenital conditions will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least twenty-five (25) years of age with hematuria, dysuria or other irritative voiding symptoms, without evidence of other causative factors such as infections or stones.

Exclusion Criteria:

* Females who are pregnant (ascertained by history)
* Females who are menstruating or within three (3) days of their last menstruation
* Patients who have undergone invasive procedures of the urogenital tract in the past two (2) months
* Patients with a history of transitional cell carcinoma (TCC) of the urinary tract

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients visiting urologist (primary care, referral, community, university or hospital).
Sampling Method: Non-Probability Sample
Enrollment: 1115 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10-01 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
Histology | Up to 1 year after cystoscopy/biopsy

SECONDARY OUTCOMES:
Cystoscopy | up to 3 months after collection
Cytology | up to 3 months after collection

CONTACTS AND LOCATIONS:
Overall Officials: Jason Trama, PhD, Study Director — Medical Diagnostic Laboratories, LLC
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

REFERENCES:
- [Background] Datta A, Adelson ME, Mogilevkin Y, Mordechai E, Sidi AA, Trama JP. Oncoprotein DEK as a tissue and urinary biomarker for bladder cancer. BMC Cancer. 2011 Jun 10;11:234. doi: 10.1186/1471-2407-11-234. PMID 21663673